CLINICAL TRIAL: NCT02907762
Title: Aorfix™ Generation IV Delivery System "IntelliFlex™" Study
Brief Title: Aorfix Intelliflex First in Human Study
Acronym: FIH-NZ
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lombard Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-07
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Endovascular; EVAR; Neck Angulation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Endovascular aneurysm repair EVAR
  Other Names: Aorfix Intelliflex

SUMMARY:
The First In Human (FIH) study is a long-term, single center, non-randomized study established by Lombard Medical, Inc. to collect "on-label" data in the clinical setting on patients undergoing endovascular repair with IntelliFlex™, the latest generation of the Aorfix™ AAA Flexible Stent Graft Delivery System, for treatment of abdominal aortic and aorto-iliac aneurysms in anatomy where the aorta in the aneurysm neck is bent through an angle between 0° and 90°.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed abdominal aortic aneurysm with indication for endovascular repair.
2. Intention to electively implant the Aorfix™ Stent Graft System with IntelliFlex™ Delivery Device.

Exclusion Criteria:

1. Do not comply with the indications for Aorfix™ in the IFU.
2. Unwillingness or inability to comply with the recommended follow-up assessments according to the standards of care of the investigative site.
3. Unwillingness or inability to provide informed consent to both the study and the EVAR procedure.
4. Patients in whom Aorfix™ is being placed as a secondary procedure to a previous surgical or endovascular treatment of an AAA other than with another Aorfix™ graft.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Diagnosed abdominal aortic aneurysm with indication for endovascular repair.
  2. Intention to electively implant the Aorfix™ Stent Graft System with IntelliFlex™ Delivery Device.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Successful Implant Delivery (30d) | 1 Month
  Successful implant delivery is also called Primary Technical Success, defined as successful introduction and deployment of the device in the absence of surgical conversion or mortality, Type I or III endoleaks, or graft limb obstruction.
  The numbers of participants having Primary Technical Success on completion of the index procedure and Clinical Success 12 months after the procedure will be recorded.
Number of participants with Treatment Success (1year) | 12 Months
  Treatment success, or Clinical Success, requires successful deployment of the endovascular device at the intended location without death as a result of aneurysm-related treatment, Type I or III endoleak, graft infection or thrombosis, aneurysm expansion (diameter >=5 mm, or volume >=5%), aneurysm rupture, or conversion to open repair.
  The numbers of participants having Primary Technical Success on completion of the index procedure and Clinical Success 12 months after the procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — University of Auckland, NZ